CLINICAL TRIAL: NCT02210364
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of Lurbinectedin (PM01183) in Combination With Capecitabine in Patients With Unresectable Metastatic Breast Cancer (MBC), Pancreatic Cancer (PC) or Metastatic Colorectal Cancer (CRC)
Brief Title: Study of Lurbinectedin (PM01183) in Combination With Capecitabine in Patients With Metastatic Breast Cancer (MBC), Pancreatic Cancer (PC) or Metastatic Colorectal Cancer (CRC).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM1183-A-006-12
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Breast Cancer; Pancreatic Cancer; Metastatic Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms | interventions — PM 01183; Capecitabine

ARMS (1):
- lurbinectedin (PM01183) and capecitabine (Experimental)
  Interventions: Drug: lurbinectedin (PM01183); Drug: capecitabine

INTERVENTIONS:
Drug: lurbinectedin (PM01183) — lurbinectedin (PM01183) 1 mg and 4 mg vials
Drug: capecitabine — capecitabine 150 mg tablets

SUMMARY:
Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of Lurbinectedin (PM01183) in Combination with Capecitabine in Patients with Unresectable Metastatic Breast Cancer (MBC), Pancreatic Cancer (PC) or Metastatic Colorectal Cancer (CRC) to determine the recommended dose (RD) of PM01183 in combination with capecitabine, to characterize the safety profile, to explore the feasibility of PM01183 dose optimization, to characterize the pharmacokinetics (PK), to obtain preliminary information on the clinical antitumor activity of this combination and to conduct an exploratory pharmacogenomic (PGx) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed and dated written informed consent (IC)
* Age between 18 and 75 years
* Women of childbearing potential must have pregnancy excluded by appropriate testing before study entry.
* Life expectancy ≥ 3 months.
* Patients with a histologically/cytologically confirmed diagnosis of unresectable Metastatic Breast Cancer, Pancreatic Cancer or metastatic Colorectal Cancer.

Exclusion Criteria:

* Three or more prior chemotherapy-containing lines for advanced disease.
* Prior treatment with PM01183 or with capecitabine containing therapy for advanced disease.
* History within the last year or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically relevant valvular heart disease or symptomatic arrhythmia or any asymptomatic ventricular arrhythmia requiring ongoing treatment.
* Ongoing chronic hepatopathy of any origin.
* Active uncontrolled infection.
* Patients with dyspnea who are requiring any ongoing oxygen support.
* Known human immunodeficiency virus (HIV) infection.
* Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
* Men or women of childbearing potential who are not using an effective method of contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Recommended dose of PM01183 in combination with capecitabine | 30 months

CONTACTS AND LOCATIONS:
Locations (2):
- Brussels, Belgium
- Barcelona, Spain